CLINICAL TRIAL: NCT07384117
Title: Long-term Outcomes of Urethral Ligament Plication and Uterosacral Ligament Plication: a Multicenter Prospective Study
Brief Title: Long-term Outcomes of Urethral and Uterosacral Ligament Plication
Acronym: ULP-USL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alev Esercan (Other Government)
Responsible Party: Sponsor-Investigator, Alev Esercan, Assoc. Prof., Sanliurfa Education and Research Hospital
Organization: Sanliurfa Education and Research Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEAH-USL/ULP
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Incontinence Stress; Incontinence, Urge
Keywords: stress urinary incontinence; urge urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary incontinent patients will have surgeries according to their incontinence type "stress" (Experimental): Urethral plication surgery (ULP) will be done for stress incontinence
  Interventions: Procedure: uterosacral ligament plication, urethral ligament plication
- Urinary incontinent patients will have surgeries according to their incontinence type "urge" (Experimental): USL for urge urinary incontinence will be done.
  Interventions: Procedure: uterosacral ligament plication, urethral ligament plication

INTERVENTIONS:
Procedure: uterosacral ligament plication, urethral ligament plication — Urethral ligament plication: With an 18-inch French Foley catheter inserted, a vertical incision of approximately 3 cm is made in the sulcus of the anterior-lateral vaginal wall, 2 cm laterally on each side of the midline, ensuring the urethral meatus remains midline. The external urethral ligaments are located inferolateral to the urethra on both sides, the urethral portion of the pubourethral ligament (PUL) is located midline, and the lateral portion of the PUL is located laterally. Using 2-0 polyester sutures, the ligaments are sutured separately on both sides to form a loop. The incised anterior vaginal tissue is then closed individually with 2-0 rapid polyglactin sutures.
  Uterosacral ligament plication: A 18F Foley catheter inserted, in the lithotomy position; the posterior cervical lip is grasped with a tenaculum, and elevated outwards and upwards. Leaving rectovaginal fascia and rectum posterior; suturing the both uterosacral ligament by 2-0 polyester sutures in the midline.

SUMMARY:
The aim of this study is to determine the long-term success and outcomes of urethral ligament plication surgeries in patients with stress incontinence and uterosacral ligament plication surgeries in patients with urge incontinence.

DETAILED DESCRIPTION:
For patients experiencing stress urinary incontinence during coughing and sneezing, which increases the intra-abdominal pressure, urethral ligament (pubourethral ligament/external urethral ligament) surgery will be performed. For patients with urge incontinence (inability to hold urine immediately) and posterior compartment syndrome (nocturia, constipation/fecal incontinence), uterosacral ligament plication surgery will be performed. For patients with both types of urinary incontinence, both surgeries will be performed, and the 2-year postoperative results will be evaluated.

This study will be a double-blind, prospective experimental study. Patients with stress urinary incontinence will undergo preoperative examination using an integral theory questionnaire to assess their symptoms and complaints anatomically and physiologically. The surgeon will always be the same person (Esercan A), and patients will be called for a follow-up examination two years after surgery (routine postoperative check-ups will be performed, but our study will focus on the results at the end of the second year). This examination will be conducted by the same surgeon, different from those who performed the surgery and published the findings, and the integral theory questionnaire will be used again for evaluation. Integral theory was defined in the literature by Professor Peter Emanuel Papa Petros from our research team, and he also provided the integral theory questionnaire. We already use this questionnaire in routine practice. Additionally, any postoperative complications will be recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over with urinary incontinence (stress or urge incontinence, or both)

  * Agreement to undergo surgery
  * No contraindications for anesthesia for surgery

Exclusion Criteria:

* Pregnancy

  * Being under 18 years of age
  * Suspicion of malignancy
  * Urinary incontinence due to neurogenic bladder
  * Presence of intrinsic sphincter (urethral) insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with urinary incontinence at any ages
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
The success (continence) rates after the operations | At postoperative first and second year
  Urinary incontinence status will be evaluated by Integral Theory Questionnaire and examinations at postoperative first and second year

SECONDARY OUTCOMES:
The complications | At second postoperative year
  Any complication seen after until postoperative second year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Emanuel Papa Petros, Prof., Study Director
Locations (1):
- Sanliurfa Education and Training Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the study will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 1 March 2026, the data will be available.
Access Criteria: Data sharing site and doi will be shared if it is asked to access.
URL: https://figshare.com/